CLINICAL TRIAL: NCT03111745
Title: Retrospective Study of Viral Reactivation Across All Bone Marrow Transplant Protocols Since 2010
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917079; 17-C-N079
Record Dates: First submitted 2017-04-12; First posted 2017-04-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08-27

CONDITIONS: Viral Infections
Keywords: Reactivation or Proliferation of Latent Viral Infections.; Viral Infection; Lymphoproliferation; Natural History
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Retrospective chart review of patients who have underwent hematopoietic stem cell transplantation (HSCT)

SUMMARY:
Background:

Some blood and immune disorders can be helped with HSCT. This is allogeneic hematopoietic stem cell transplantation. The person who gets the stem cells has their immune system suppressed. This is done to help prevent their body from rejecting the transplant. During this time, the person is at a high risk to get viral infections. Researchers want to study the records of people who had transplants a few years ago. They want to look at how often certain viral complications happened.

Objective:

To study how often certain viral complications occurred after HSCT and what risks factors were involved.

Eligibility:

Records will be reviewed. No participants will be contacted.

Design:

Researchers will review medical records from the NIH Clinical Center.

The records will be from people who had HSCT between 2010 and 2015 when they were between 4 and 85 years old. They already gave consent for their data to be studied.

Data collected will include:

Vital statistics like age and sex

Viral status of the recipient and donor

Reason for transplant

Transplant details

How the immune system recovered after transplant

If the recipient got graft versus host disease

Any infections

Overall survival

DETAILED DESCRIPTION:
This protocol is a retrospective chart review of patients who have underwent hematopoietic stem cell transplantation (HSCT) at the NIH Clinical Center. If this proposal is approved, BTRIS will identify and populate the patients in these protocols, and BTRIS identified reports will be used going forward.

BTRIS identified reports will be used to review patient progress notes, all aspects of the transplant platform, as well as viral titers over the course of each patient s follow-up, supplemented by review of paper or CRIS electronic medical records as needed.

The study will involve review of patient records and will not use specimens or participant contact. The participants whose records will be reviewed in this protocol were enrolled in NIH protocols between 2010 and December 1, 2020. BTRIS policy requires approval from Principal Investigators on certain protocols. These Principal Investigators have been contacted via email for permission to conduct this study and have verified that none of the original protocols or informed consent documents precludes such a review of clinical data.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Subjects will not be recruited for this study.

Ages: 4 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This protocol is a retrospective chart review of patients who have underwent hematopoietic stem cell transplantation (HSCT) at the NIH Clinical Center
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2018-12-29 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
To determine the incidence and risk factors for various viral complications by HSCT platform and its relation to immune reconstitution. | 1 year
  Incidence and risk factors for various viral complications by HSCT platform and its relation to immune reconstitution.

SECONDARY OUTCOMES:
incidence of late CMV, EBV, BK cystitis, adenovirus, HHV6 encephalitis, JC virus, and CNS disease | 1 year
  incidence of late CMV, EBV, BK cystitis, adenovirus, HHV6 encephalitis, JC virus, and CNS disease
Evaluate the relationship between EBV and CMV in blood | 1 year
  Evaluate the relationship between EBV and CMV in blood
evaluate relationship between viral infection and immunologic parameters | 1 year
  evaluate relationship between viral infection and immunologic parameters
evaluate relationship between GVHD and viral infection incidence/burden | 1 year
  evaluate relationship between GVHD and viral infection incidence/burden
determine overall survival and incidence of infection-related mortality | 1 year
  determine overall survival and incidence of infection-related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dimana Dimitrova, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Tischer J, Engel N, Fritsch S, Prevalsek D, Hubmann M, Schulz C, Zoellner AK, Bucklein V, Reibke R, Mumm F, Rieger CT, Hill W, Ledderose G, Stemmler HJ, Kohnke T, Jager G, Kolb HJ, Schmid C, Moosmann A, Hausmann A. Virus infection in HLA-haploidentical hematopoietic stem cell transplantation: incidence in the context of immune recovery in two different transplantation settings. Ann Hematol. 2015 Oct;94(10):1677-88. doi: 10.1007/s00277-015-2423-y. Epub 2015 Jun 10. PMID 26055139
- [Background] Kang E, Gennery A. Hematopoietic stem cell transplantation for primary immunodeficiencies. Hematol Oncol Clin North Am. 2014 Dec;28(6):1157-70. doi: 10.1016/j.hoc.2014.08.006. Epub 2014 Sep 16. PMID 25459185
- [Background] Reddehase MJ. Mutual Interference between Cytomegalovirus and Reconstitution of Protective Immunity after Hematopoietic Cell Transplantation. Front Immunol. 2016 Aug 4;7:294. doi: 10.3389/fimmu.2016.00294. eCollection 2016. PMID 27540380